CLINICAL TRIAL: NCT00827593
Title: Managing Obesity by Combining Behavioral Weight Loss and Commercial Approaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baruch College City University of New York (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Angela M Pinto, Assistant Professor of Psychology, Baruch College City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070601
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard behavioral weight loss (Active Comparator): University-based behavioral weight loss treatment
  Interventions: Behavioral: Standard behavioral weight loss treatment
- Weight Watchers (Active Comparator): Weight Watchers program
  Interventions: Behavioral: Weight Watchers
- Combined Treatment (Active Comparator): University-based behavioral weight loss treatment followed by Weight Watchers
  Interventions: Behavioral: Combined Treatment

INTERVENTIONS:
Behavioral: Standard behavioral weight loss treatment — Participants will receive 12 months of university-based behavioral weight loss treatment
  Arms: Standard behavioral weight loss
Behavioral: Weight Watchers — Participants will receive 12 months of Weight Watchers
  Arms: Weight Watchers
Behavioral: Combined Treatment — Participants will receive university-based behavioral weight loss treatment followed by Weight Watchers
  Arms: Combined Treatment

SUMMARY:
The purpose of this study is to examine the effectiveness of 3 behavioral weight loss programs- Weight Watchers, university-based behavioral weight loss treatment, and a combined approach which includes university-based treatment followed by Weight Watchers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30-65 years
* BMI between 27-50 kg/m2
* Written approval/consent from primary health care provider

Exclusion Criteria:

* Unable to walk 2 blocks without stopping.
* Currently participating in a weight loss program or taking weight loss medication.
* Participated in a weight loss program in the last year
* Took weight loss medication in the last 6 months.
* Participated in Weight Watchers in last 2 years.
* Lost >=5% of body weight during 6 months prior to screening.
* Pregnant, lactating, less than 6 months postpartum, or plan to become pregnant during study time frame.
* Report conditions that in the judgment of the principal investigator would render them potentially unlikely to follow protocol for the 12 month study.
* Report a medical condition that would affect the safety and/or efficacy of a weight management program involving changes in diet and physical activity.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
weight loss | 3, 6, 12 months

SECONDARY OUTCOMES:
cost-effectiveness | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Pinto, PhD, Principal Investigator — Baruch College
Locations (1):
- Baruch College, New York, New York, United States

REFERENCES:
- [Derived] Pinto AM, Fava JL, Hoffmann DA, Wing RR. Combining behavioral weight loss treatment and a commercial program: a randomized clinical trial. Obesity (Silver Spring). 2013 Apr;21(4):673-80. doi: 10.1002/oby.20044. PMID 23404824